CLINICAL TRIAL: NCT00680199
Title: Information Processing at Sleep Onset and During Sleep in Patients With Insomnia
Acronym: COTE
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sara Matteson, Clinical Assistant Professor, University of Rochester
Other Study IDs: RSRB # 20615; R21MH076855 (NIH)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Primary Insomnia
Keywords: Insomnia; Primary Insomnia; Good Sleepers; ERP
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Primary Insomnia
- 2: Good Sleepers

SUMMARY:
Chronic insomnia is thought to occur as a result of hyperarousal. While there is a wealth of data to support this position, there is a lack of research to define how hyperarousal interferes with sleep initiation, maintenance, and the perception of sleep quality and quantity. We propose to use Event-related Potential (ERP) techniques to evaluate information processing at sleep onset and during sleep. ERP measures of information processing have been well established in good sleepers; they have not been, however, applied to the problem of insomnia. The goal of the project is to examine the premise that the occurrence and severity of insomnia is fundamentally related to a neurobiologic preparedness to "attend to" and "identify" environmental stimuli. Following an extensive screening, patients with insomnia and good sleepers will participate in two experimental conditions, requiring that they spend four nights in the sleep laboratory over a two week period. ERP data will be gathered prior to, following, and during sleep.

The ultimate objectives for this line of research are to determine 1) if insomnia is associated with a failure to inhibit information processing at sleep onset and/or during sleep, 2) if the failure to inhibit information processing at sleep onset and/or during sleep is associated with the occurrence and/or severity of insomnia symptoms, 3) what brain regions are functioning differently so as to give rise to information processing abnormalities, and 4) the extent to which pharmacologic and/or Cognitive Behavioral treatment for insomnia alters information processing abnormalities and/or the associated brain activity.

ELIGIBILITY:
Inclusion Criteria for Psychophysiologic Insomnia (PI)

These subjects will meet RDC criteria for Psychophysiologic insomnia. In addition, the complaint of disturbed sleep will have at least one of the following minimal characteristics:

* > 30 min. sleep-onset latency (SL) (Initial Insomnia)
* >2 awakenings per night (>15 min. ea.) and/or wake after sleep-onset (WASO) of > 30 min (Middle Insomnia)

Total Sleep Time (TST) will not exceed 6 hours [unless the Sleep Efficiency (SE) quotient is < 80%] and the problem frequency must be > 4 nights/week (Severe Insomnia) with a problem duration > 6 months (Chronic Insomnia)B .

Inclusion Criteria for Good Sleeper Subjects

* Report that they obtain enough sleep and that their sleep is restorative
* Have a score of less than 10 on the Epworth Sleepiness Scale (ESS)50-52
* Have a score of less than 15 on the Ford Insomnia Response to Stress Test (FIRST)53
* Have a score of less than 7 on the Insomnia Severity Index (ISI)54
* Report retrospectively and prospectively < 15 minutes to fall asleep and "wake after sleep onset time" of < 15 minutes and a total sleep time > 6 hoursA

A These profiles will be evident at both intake (based on retrospective reports) and as an average from the two weeks of baseline diaries (based on prospective sampling).

Exclusion Criteria for All Subjects

• Unstable medical illness or acute or history of psychiatric illness (except GAD or MDD - Allowed provided that these have resolved and not recurred within 5 years) As ascertained with self report questionnaires, a clinical History, a physical exam and a clinical chemistry profile.

To assure that the insomnia is not secondary to these factors

* Symptoms suggestive of sleep disorders other than insomnia To assure that the insomnia is not secondary to these factors
* Polysomnographic data indicating sleep disorders other than insomnia To assure that the insomnia is not secondary to these factors
* History of head injury with a sustained loss of consciousness To help assure that the EEG measures are unconfounded by brain damage
* Evidence of active illicit substance use or fitting criteria for alcohol abuse or dependence To assure that the insomnia is not secondary to these factors
* Use of CNS active medications including antidepressants and hypnotics (within 2 weeks or 5 half-lives) To help assure that the EEG measures are unconfounded by medication effects such as the "BZ artifact".
* Inadequate language comprehension To assure the quality of self report data as all the measures are in English.
* Pregnancy Excluded owing to the hormonal changes that occur with pregnancy
* Left Handedness To control for EEG differences related to handedness
* Nicotine Use To assure that the insomnia is not secondary to these factors
* Caffeine use that exceeds 2 beverages per day or occurs past 5pm in the evening.

To assure that the insomnia is not secondary to these factors

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The intent of this study is to assess whether patients with insomnia exhibit an increased level of information processing (as assessed with ERP methods) at sleep onset and during polysomnographically defined sleep. | 2 years

SECONDARY OUTCOMES:
Assess spindle and K-complex density to investigate whether the groups differ with respect to these putative markers of information processing and parse ERP trials in NREM into those with and without spindles and K-complexes in order to investigate their | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara E Matteson-Rusby, Psy.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Sleep and Neurophysiology Research Lab, Rochester, New York, United States